CLINICAL TRIAL: NCT02357511
Title: Validation of Pulse Waveform Analysis-based Continuous Noninvasive Blood Pressure Measurement Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MEDIETA2015
Record Dates: First submitted 2015-01-22; First posted 2015-02-06 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Blood Pressure
Keywords: sensitivity; specificity; novel blood pressure monitor; Saturation
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study goup (Experimental): Vital values are being measured for the time of two hours at postoperative setting at postanesthesia care unit. A novel method is compared to golden standard: invasive measurement. Also Saturation measurements are being compared between standard and study monitor.
  Interventions: Device: Study Monitor used

INTERVENTIONS:
Device: Study Monitor used

SUMMARY:
The study aims to define the sensitivity and specificity of a novel continuous noninvasive blood pressure monitor.

DETAILED DESCRIPTION:
A novel continuous noninvasive blood pressure monitor is compared to invasive arterial measurement at postoperative care unit after a planned operation. Monitor captures also saturation and ECG, which are compared to traditional monitoring.

ELIGIBILITY:
Inclusion Criteria:

* subjected to operative treatment with the need for invasive blood pressure measurement
* spontaneous ventilation
* able to give informed consent

Exclusion Criteria:

* denial by patient
* pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Relationship between invasive and noninvasive blood pressure measurement | 2 hours of continuous measurement at PACU
  comparability of study monitor systolic, diastolic and mean blood pressure to invasive blood pressure measurement

SECONDARY OUTCOMES:
Relationship between study monitor Sp02 measurement and current sp02 measurement | 2 hours of continuous measurement at PACU
  comparability of measurements at several timepoints recorded as 10s intervals

CONTACTS AND LOCATIONS:
Overall Officials: Arvi Yli-Hankala, Professor, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland